CLINICAL TRIAL: NCT04558008
Title: Effectiveness of Online Mindfulness-based Stress Reduction Among Teachers at Upper Secondary Schools and Schools of Health and Social Care
Brief Title: Effectiveness of MBSR Among Teachers at Upper Secondary Schools and Schools of Health and Social Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 07072020
Record Dates: First submitted 2020-09-16; First posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-07

CONDITIONS: Stress Reduction; Mental Well-being
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online MBSR (Experimental): MBSR according to international standards (2.5 hours group session once a week in 8 weeks; a silence retreat day; and 45-60 minutes homework six days a week). Content in accordance with MBSR curriculum.
  Interventions: Behavioral: Online MBSR
- Wait-list control (No Intervention): Usual practice

INTERVENTIONS:
Behavioral: Online MBSR — Described previously
  Arms: Online MBSR

SUMMARY:
The aim is to evaluate the effectiveness of online Mindfulness-based Stress Reduction among school teachers in Danish upper secondary schools and schools of health and social care on mental well-being in the teachers and their students. The study is a cluster-randomised trial including 43 schools; 76 teachers; 1.000 students.

ELIGIBILITY:
Inclusion Criteria:

* School teacher at a Danish upper secondary school or school of health and social care that commit to participate in a trial aiming to implement and evaluate the effectiveness of a school-based mindfulness programme.

Exclusion Criteria:

* acute treatment-demanding clinical depression or a diagnosis of psychosis or schizophrenia
* abuse of alcohol, drugs, medicine

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2021-10-28 (Estimated); Study Completion 2021-10-28 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale | 6 months from baseline
  Change in perceived stress among the school teachers

SECONDARY OUTCOMES:
Perceived Stress Scale | post MBSR (8 weeks from baseline) and 12 months from baseline
  Change in perceived stress among the school teachers
Brief Resilience Scale | post MBSR (8 weeks from baseline), 6 and 12 months from baseline
  Change in resilience among the school teachers
Symptom Check List - 5 | post MBSR (8 weeks from baseline), 6 and 12 months from baseline
  Change in symptoms of anxiety and depression among the school teachers
WHO-5 | post MBSR (8 weeks from baseline), 6 and 12 months from baseline
  Change in well-being among the school teachers
Five Facet Mindfulness Questionnaire-15 | post MBSR (8 weeks from baseline), 6 and 12 months from baseline
  Change in mindfulness among the school teachers
Amsterdam Resting State Questionnaire | post MBSR (8 weeks from baseline), 6 and 12 months from baseline
  Change in resting state among the school teachers

CONTACTS AND LOCATIONS:
Overall Officials: Lone Fjorback, PhD, MD, Study Director — Aarhus University, Danish Center for Mindfulness
Locations (1):
- Danish Center for Mindfulness, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Individual deidentified participant data will be shared by reasonable request, following publication of planned papers.
Supporting Information: Study Protocol, SAP